CLINICAL TRIAL: NCT02937012
Title: Efficacy and Security of Bezafibrate in Patients With Primary Biliary Cirrhosis Without Biochemical Response to Ursodeoxycholic Acid: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Use of Bezafibrate in Patients With Primary Biliary Cirrhosis to Archive Complete Biochemical Response in Non-responders
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Eric Lopez Mendez, Hepatologist, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1757
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cirrhosis; Primary Biliary Cholangitis; Bezafibrate; Ursodeoxycholic acid
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Bezafibrate; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bezafibrate & Ursodeoxycholic acid (Experimental): Bezafibrate 200 mg capsule every 12 hours and ursodeoxycholic acid at a dose of 13 to 15 mg per Kg per day, for 12 months
  Interventions: Drug: Bezafibrate; Drug: Ursodeoxycholic Acid
- Placebo & Ursodeoxycholic acid (Placebo Comparator): Placebo capsule (for bezafibrate 200 mg capsule) every 12 hours and ursodeoxycholic acid at a dose of 13 to 15 mg per Kg per day, for 12 months
  Interventions: Drug: Ursodeoxycholic Acid; Drug: Placebo (for Bezafibrate)

INTERVENTIONS:
Drug: Bezafibrate — Bezafibrate 200 mg manufactured in a pill/capsule presentation
  Other Names: Bezalip
  Arms: Bezafibrate & Ursodeoxycholic acid
Drug: Ursodeoxycholic Acid — The patients will continue with the administration of ursodeoxycholic acid at a dose of 13 to 15 mg per Kg per day throughout the study
  Other Names: Ursofalk
Drug: Placebo (for Bezafibrate) — Starch pill/capsule manufactured to mimic bezafibrate 200 mg tablet
  Other Names: Does not apply
  Arms: Placebo & Ursodeoxycholic acid

SUMMARY:
The primary biliary cholangitis (PBC), formerly known as primary biliary cirrhosis, treatment is based in the use of ursodeoxycholic acid (UDCA) at a daily dose of 13 to 15 mg/kg, without other treatment options. Patients with good or complete response to UDCA have more liver transplant-free survival and delay histologic progression compared to patients with partial or no response. Nowadays there is an estimated partial response to UDCA in approximately 30 to 50% of patients with PBC. There is a need for new second line management strategies for patients without a biochemical response to UDCA.

The addition of bezafibrate to the treatment of PBC patients with partial biochemical response to UDCA, will increase the biochemical response and improve the long term prognosis? And if so, which are the efficacy and security of bezafibrate in PBC patients without biochemical response?

DETAILED DESCRIPTION:
There are case reports and pilot studies in patients with primary biliary cholangitis (PBC) In the literature in which the effect of fibrates (specially bezafibrate) on the improvement of biochemical cholestasis have been seen, however the clinical benefit (survival, mortality, fatigue, pruritus) has not been reported and likewise the response criteria used in previous studies is very heterogeneous. In previous studies, bezafibrate has been proved to be a secure drug in this patients, with few adverse events, also it is an economic and of easy access drug. For all this the investigators intent to study the utility of bezafibrate as an additional treatment in PBC patients without response to UDCA.

This is a randomized, placebo-controlled, parallel-group study designed to enroll a total of 34 patients with diagnosis of PBC without a complete response to the use of UDCA for more than a year, then the participants will be divided by randomization to receive bezafibrate or placebo, resulting in a total of two groups of 17 patients each. Both groups will be followed every 3 months for a total of 1 year with clinical and laboratory follow-up to determine the efficacy and security of the treatment. The investigators will measure all the laboratory variables related to the disease and possible adverse effects of the use of fibrates (creatine kinase, transaminases, bilirubin, alkaline phosphatase), also the investigators will measure the quality of life variables (pruritus severity, Short Form [SF]-36 questionnaire), and determine the fibrosis stage at the beginning and end of the study by non-invasive methods (transient elastography).

The study is directed to patients with PBC diagnosis who have had management with standard UDCA dose (13 to 15 mg/kg per day) for at least 6 months and had not reached complete biochemical response, defined by Paris II criteria. The dose of fibrate to use will be bezafibrate 200 mg every 12 hours or placebo every 12 hours for 12 months, both having the exact characteristics to avoid their recognition. Patients will continue the administration of UDCA at the same dose at enrollment. The intervention will be for a period of 12 months, with a follow-up every 3 months completing 5 medical follow-up visits (0, 3, 6, 9 and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Primary biliary cirrhosis diagnosis made by 2 of the 3 criteria:

  1. Biochemical evidence of cholestasis with an alkaline phosphatase rise of 1.5 times the upper normal limit.
  2. Anti-mitochondrial antibodies positivity
  3. Histopathologic evidence of a nonsuppurative cholangitis and small bile ducts destruction
* Use of ursodeoxycholic acid (UDCA) for at least 6 months at enrollment at a therapeutic dose (13 to 15 mg per Kg per day)
* Evidence of a suboptimal biochemical response to UDCA, defined by the presence of one of the Paris II criteria:

  1. Alkaline phosphatase more or equal to 1.5 times the normal upper limit
  2. Aspartate transaminase more or equal to 1.5 times the normal upper limit
  3. Bilirubin more than 1 mg/dL
* Signed informed consent.

Exclusion Criteria:

* No informed consent given to enrollment
* Actual or history of hepatic decompensation (ascitis, variceal upper gastrointestinal bleeding, hepatic encephalopathy)
* Secondary immunosuppression caused by drugs (for example; steroids), use of statins or fibrates in the last 6 months. The investigators will exclude patients with medical indication of statin use.
* Coexistence of hepatopathy, chronic viral infections like C hepatitis virus, B virus and HIV. Excessive alcohol intake, autoimmune hepatitis, non-alcoholic fatty liver disease (diagnosed by histopathology), Wilson disease, hemochromatosis, celiac disease, choledocolithiasis, non-controlled thyroid disease
* Post liver transplant
* Known allergy or intolerance to fibrates
* Pregnancy or women who desire to become pregnant
* Chronic kidney disease with a glomerular filtration less than 60 ml/min
* Patients under total anticoagulation with vitamin K antagonist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Complete biochemical response | 12 months
  The complete biochemical response in patients with primary biliary cholangitis is defined as the reduction of alkaline phosphatase lower than 1.5 times the upper normal limit, reduction of aspartate transaminase lower than 1.5 times the upper normal limit and bilirubin lower than 1 mg/dL

SECONDARY OUTCOMES:
Increase in liver transaminases or development of rhabdomyolysis | Follow-up every 3 months for 12 months.
  Elevation of transaminases of biochemical evidence of rhabdomyolysis.

OTHER OUTCOMES:
Comparison of fatigue between groups | Two evaluations: At enrollment and 12 months later.
  Clinical evaluation of fatigue with the use of the Krupp´s Fatigue Severity Scale.
Quality of life | Two evaluations: At enrollment and 12 months later.
  Evaluation of the quality of life with the SF-36 questionnaire.
Pruritus intensity | Follow-up every 3 months for 12 months.
  Evaluation made by the use of visual analogue scales.
Liver fibrosis evaluation by a non-invasive method | Two evaluations: At enrollment and 12 months later.
  Evaluation of the liver fibrosis by transient elastography.
Disease natural history outcome | Two evaluations: At enrollment and 12 months later.
  Compare the liver transplant-free survival, overall survival and liver decompensation-free survival between groups.
Prognostic scales comparison | Two evaluations: At enrollment and 12 months later.
  Compare the different prognostic scales (Mayo, Child-Pugh and MELD) between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Edgardo Eric Lopez Mendez, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Flores A, Mayo MJ. Primary biliary cirrhosis in 2014. Curr Opin Gastroenterol. 2014 May;30(3):245-52. doi: 10.1097/MOG.0000000000000058. PMID 24671010
- [Result] Lindor KD, Gershwin ME, Poupon R, Kaplan M, Bergasa NV, Heathcote EJ; American Association for Study of Liver Diseases. Primary biliary cirrhosis. Hepatology. 2009 Jul;50(1):291-308. doi: 10.1002/hep.22906. No abstract available. PMID 19554543
- [Result] Selmi C, Invernizzi P, Keeffe EB, Coppel RL, Podda M, Rossaro L, Ansari AA, Gershwin ME. Epidemiology and pathogenesis of primary biliary cirrhosis. J Clin Gastroenterol. 2004 Mar;38(3):264-71. doi: 10.1097/00004836-200403000-00013. PMID 15128074
- [Result] Boonstra K, Beuers U, Ponsioen CY. Epidemiology of primary sclerosing cholangitis and primary biliary cirrhosis: a systematic review. J Hepatol. 2012 May;56(5):1181-1188. doi: 10.1016/j.jhep.2011.10.025. Epub 2012 Jan 13. PMID 22245904
- [Result] Jones DE, Bhala N, Burt J, Goldblatt J, Prince M, Newton JL. Four year follow up of fatigue in a geographically defined primary biliary cirrhosis patient cohort. Gut. 2006 Apr;55(4):536-41. doi: 10.1136/gut.2005.080317. Epub 2005 Nov 18. PMID 16299032
- [Result] van Os E, van den Broek WW, Mulder PG, ter Borg PC, Bruijn JA, van Buuren HR. Depression in patients with primary biliary cirrhosis and primary sclerosing cholangitis. J Hepatol. 2007 Jun;46(6):1099-103. doi: 10.1016/j.jhep.2007.01.036. Epub 2007 Mar 2. PMID 17399846
- [Result] Talwalkar JA, Souto E, Jorgensen RA, Lindor KD. Natural history of pruritus in primary biliary cirrhosis. Clin Gastroenterol Hepatol. 2003 Jul;1(4):297-302. PMID 15017671
- [Result] Prince M, Chetwynd A, Newman W, Metcalf JV, James OF. Survival and symptom progression in a geographically based cohort of patients with primary biliary cirrhosis: follow-up for up to 28 years. Gastroenterology. 2002 Oct;123(4):1044-51. doi: 10.1053/gast.2002.36027. PMID 12360466
- [Result] Springer J, Cauch-Dudek K, O'Rourke K, Wanless IR, Heathcote EJ. Asymptomatic primary biliary cirrhosis: a study of its natural history and prognosis. Am J Gastroenterol. 1999 Jan;94(1):47-53. doi: 10.1111/j.1572-0241.1999.00770.x. PMID 9934730
- [Result] Shi J, Wu C, Lin Y, Chen YX, Zhu L, Xie WF. Long-term effects of mid-dose ursodeoxycholic acid in primary biliary cirrhosis: a meta-analysis of randomized controlled trials. Am J Gastroenterol. 2006 Jul;101(7):1529-38. doi: 10.1111/j.1572-0241.2006.00634.x. PMID 16863557
- [Result] Poupon RE, Bonnand AM, Chretien Y, Poupon R. Ten-year survival in ursodeoxycholic acid-treated patients with primary biliary cirrhosis. The UDCA-PBC Study Group. Hepatology. 1999 Jun;29(6):1668-71. doi: 10.1002/hep.510290603. PMID 10347106
- [Result] ter Borg PC, Schalm SW, Hansen BE, van Buuren HR; Dutch PBC Study Group. Prognosis of ursodeoxycholic Acid-treated patients with primary biliary cirrhosis. Results of a 10-yr cohort study involving 297 patients. Am J Gastroenterol. 2006 Sep;101(9):2044-50. doi: 10.1111/j.1572-0241.2006.00699.x. Epub 2006 Jul 18. PMID 16848809
- [Result] Pares A, Caballeria L, Rodes J. Excellent long-term survival in patients with primary biliary cirrhosis and biochemical response to ursodeoxycholic Acid. Gastroenterology. 2006 Mar;130(3):715-20. doi: 10.1053/j.gastro.2005.12.029. PMID 16530513
- [Result] Angulo P, Batts KP, Therneau TM, Jorgensen RA, Dickson ER, Lindor KD. Long-term ursodeoxycholic acid delays histological progression in primary biliary cirrhosis. Hepatology. 1999 Mar;29(3):644-7. doi: 10.1002/hep.510290301. PMID 10051462
- [Result] Corpechot C. Primary biliary cirrhosis and bile acids. Clin Res Hepatol Gastroenterol. 2012 Sep;36 Suppl 1:S13-20. doi: 10.1016/S2210-7401(12)70016-5. PMID 23141888
- [Result] Corpechot C, Abenavoli L, Rabahi N, Chretien Y, Andreani T, Johanet C, Chazouilleres O, Poupon R. Biochemical response to ursodeoxycholic acid and long-term prognosis in primary biliary cirrhosis. Hepatology. 2008 Sep;48(3):871-7. doi: 10.1002/hep.22428. PMID 18752324
- [Result] Corpechot C, Carrat F, Poujol-Robert A, Gaouar F, Wendum D, Chazouilleres O, Poupon R. Noninvasive elastography-based assessment of liver fibrosis progression and prognosis in primary biliary cirrhosis. Hepatology. 2012 Jul;56(1):198-208. doi: 10.1002/hep.25599. Epub 2012 Jun 5. PMID 22271046
- [Result] Honda A, Ikegami T, Nakamuta M, Miyazaki T, Iwamoto J, Hirayama T, Saito Y, Takikawa H, Imawari M, Matsuzaki Y. Anticholestatic effects of bezafibrate in patients with primary biliary cirrhosis treated with ursodeoxycholic acid. Hepatology. 2013 May;57(5):1931-41. doi: 10.1002/hep.26018. Epub 2013 Apr 5. PMID 22911624
- [Result] Cuperus FJ, Halilbasic E, Trauner M. Fibrate treatment for primary biliary cirrhosis. Curr Opin Gastroenterol. 2014 May;30(3):279-86. doi: 10.1097/MOG.0000000000000056. PMID 24625898
- [Result] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Result] Zuniga MA, Carrillo-Jimenez GT, Fos PJ, Gandek B, Medina-Moreno MR. [Evaluation of health status using Survey SF-36: preliminary results in Mexico]. Salud Publica Mex. 1999 Mar-Apr;41(2):110-8. Spanish. PMID 10343514
- [Result] Duran-Arenas L, Gallegos-Carrillo K, Salinas-Escudero G, Martinez-Salgado H. [Towards a Mexican normative standard for measurement of the short format 36 health-related quality of life instrument]. Salud Publica Mex. 2004 Jul-Aug;46(4):306-15. doi: 10.1590/s0036-36342004000400005. Spanish. PMID 15468571
- [Result] Rudic JS, Poropat G, Krstic MN, Bjelakovic G, Gluud C. Bezafibrate for primary biliary cirrhosis. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD009145. doi: 10.1002/14651858.CD009145.pub2. PMID 22259000
- See also: Krupp´s Fatigue Severity Scale taken from the article: Valencia-Flores, et al. Sleep, Fatigue, Depression, and Pain in Mexican Women with Systemic Lupus Erythematosus: An Exploratory Study. Hisp Health Care Int. 2010 — http://www.ingentaconnect.com/contentone/springer/hhci/2010/00000008/00000004/art00006